CLINICAL TRIAL: NCT03606070
Title: Multiparametric PET-MRI Integration for a New Approach to Tumor Heterogeneity in Non-Small Cell Lung Cancer (NSCLC): Pilot Study
Acronym: IMAHTEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-A02074-47; 2016/2499 (Other: CSET number)
Record Dates: First submitted 2018-07-20; First posted 2018-07-30 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: NSCLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with NSCLC (Other): Characterization of tumor heterogeneity by multiparametric regional mapping PET-MRI.
  Patients will realize:
  * a PET-MRI examination performed before the chemoradiotherapy treatment (so-called baseline PET-MRI)
  * a PET-MRI examination performed midway through treatment (PET-MRI1 under treatment), after receiving 33 ± 4 Gy (approximately 2.5 months after the first PET-MRI).
  Interventions: Diagnostic Test: PET-MRI

INTERVENTIONS:
Diagnostic Test: PET-MRI — * a PET-MRI examination performed before the chemoradiotherapy treatment (so-called baseline PET-MRI)
  * a PET-MRI examination performed midway through treatment (PET-MRI1 under treatment), after receiving 33 ± 4 Gy (approximately 2.5 months after the first PET-MRI).

SUMMARY:
To estimate the intra and inter-operator reproducibility of multiparametric regional PET-MRI mapping in locally advanced and trace mestastatic non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced NSCLC (stages IIB, IIIA or IIIB of the TNM classification 7th edition) or trace metastatic stage IV (</=5 mestastasis, </= 3 organ reached)
2. Exclusive therapeutic management by concomitant radio-chemotherapy administered in accordance with international recommendations (dual therapy with platinum salts)
3. Signed consent
4. Patients affiliated with the social security scheme or beneficiary of a similar scheme.

Exclusion Criteria:

1. Minor
2. Pregnant / lactating woman
3. Person deprived of liberty by judicial or administrative decision, adults who are the subject of a legal protection measure or unable to express their consent
4. Previous cancer in the 2 years prior to registration
5. Previousradiotherapy / thoracic surgery
6. Patients under experimental treatment or for whom the administration of an experimental treatment is planned
7. Claustrophobic patients
8. Severe Renal Insufficiency (Clearance MDRD Cockroft <30ml / min)
9. Uncontrolled diabetes, hyperglycemia> 1.8g / L
10. Patient with metallic implants not compatible with MRI or any immovable implanted electronic medical device (eg pacemaker, neurostimulator, cochlear implants, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-11-25 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Measurement of intra and inter-operator reproducibility of multiparametric regional PET-MRI mapping performed before and under treatment. | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No